CLINICAL TRIAL: NCT07235527
Title: Real-World Outcomes of Aflibercept Biosimilar MY-1701P Treatment in Exudative Age-Related Macular Degeneration
Brief Title: Real-Life Clinical Outcomes of Aflibercept Biosimilar MY-1701P in the Treatment of Exudative Age-Related Macular Degeneration
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sinan KALPAKOĞLU, MD, Ophthalmology Consultant, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: skalpakoglu
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Age Related Macular Degeneration; Exudative Age-Related Macular Degeneration; Anti Vascular Endothelial Growth Factor
Keywords: age related macular degeneration; anti vascular endothelial growth factor; anti-VEGF; aflibercept; macular neovascularization; aflibercept biosimilar
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- patients treated with Yesafili: aflibercept biosimilar used
  Interventions: Drug: Aflibercept biosimilar (MY-1701P)

INTERVENTIONS:
Drug: Aflibercept biosimilar (MY-1701P) — Patients receiving the aflibercept biosimilar MY-1701P (marketed as Yesafili®) as part of routine clinical care.

SUMMARY:
In this study, patients receiving Eylea treatment will be treated with Yesafili, a biosimilar molecule, and routine examination results will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 45 and 90 years with active neovascular age-related macular degeneration (nAMD)
* who show signs of disease activity on routine ophthalmologic examination and optical coherence tomography (OCT)
* for whom intravitreal injection has already been clinically indicated

Exclusion Criteria:

* Patients younger than 45 years or older than 90 years
* History of stroke, cerebrovascular event, myocardial infarction, or coronary stent placement within the last six months
* Presence of uveitis
* Media opacity preventing adequate retinal imaging (e.g., corneal opacity, mature cataract)
* Coexistence of other retinal vascular diseases (e.g., branch retinal vein occlusion, diabetic macular edema)
* Presence of hereditary retinal dystrophies
* Presence of optic atrophy

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 45 to 90 years diagnosed with active neovascular (exudative) age-related macular degeneration (nAMD), who are receiving routine ophthalmologic follow-up at a tertiary referral center and have been clinically indicated for intravitreal aflibercept biosimilar (MY-1701P) injection. Participants will be selected based on evidence of disease activity on ophthalmologic examination and optical coherence tomography (OCT) imaging.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) and Central Macular Thickness After MY-1701P Injection | Baseline to Month 6
  Evaluation of anatomical and functional outcomes following intravitreal MY-1701P (aflibercept biosimilar) treatment, including presence or resolution of intraretinal and subretinal fluid, changes in central macular thickness, and improvement in best-corrected visual acuity (BCVA) measured by standardized ETDRS (Early Treatment Diabetic Retinopathy Study) or Snellen methods.

SECONDARY OUTCOMES:
Effect of MY-1701P on Pigment Epithelial Detachment, Neovascularization Size, and Treatment Interval Adjustment | Baseline to Month 6
  Assessment of the influence of MY-1701P treatment on pigment epithelial detachment (PED) height and area, macular neovascularization size, and changes in treatment intervals over the follow-up period, based on optical coherence tomography (OCT) and fluorescein angiography findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, şişli, Turkey (Türkiye)